CLINICAL TRIAL: NCT02714101
Title: Effects of Hippotherapy on the Motivation and Social Interaction/Social Communication of Children With Autism
Brief Title: Equine-assisted Occupational Therapy for Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00031008
Record Dates: First submitted 2016-03-06; First posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Equine assisted occupational therapy (Experimental): Intervention was one 40 to 60 minute session per week. Half of the session was spent riding a horse and half was spent doing horse related activities. Children had 9 to 12 sessions
  Interventions: Other: Equine assisted occupational therapy

INTERVENTIONS:
Other: Equine assisted occupational therapy — Intervention was one 40 to 60 minute session per week. Half of the session was spent riding a horse and half was spent doing horse related activities. Children had 9 to 12 sessions

SUMMARY:
Children with Autism Spectrum Disorder have difficulty engaging in activities. This study examined the effects of equine-assisted occupational therapy for 7 children with ASD ages 4 to 8 years. A multiple baseline design was used. For each child, there were 9 to 11 baseline assessments, 9 to 12 intervention sessions, and 4 follow-up sessions.

DETAILED DESCRIPTION:
Children with Autism Spectrum Disorder (ASD) have difficulty engaging in activities. Based on the literature, the unique features of horses may be beneficial to children with ASD. There is limited research supporting the use of horses in occupational therapy interventions. This study examined the effects of equine-assisted occupational therapy for 7 children with ASD ages 4 to 8 years. A multiple baseline design was used. For each child, there were 9 to 11 baseline assessments (gross and fine motor play activities), 9 to 12 intervention sessions, and 4 follow-up sessions (gross and fine motor play activities). Intervention sessions were 40 to 60 minutes long and consisted of time spent on the horse and in horse related activities. Children were videorecorded in all conditions. Trained coders scored randomly selected segments of the video recording. Inter-rater reliability was good.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Autism spectrum disorder by a multidisciplinary team,
* between ages 3 and 8,
* understand basic English,
* willing to ride a horse, no horse riding in the past 3 months.

Exclusion Criteria:

* severe of repeated aggressive behaviour,
* comorbidities such as deafness that would interfere with intervention.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Rater coding of engagement | One 5 minute segment per session for five months
  Trained coders rated the proportion of time the child was engaged in the activities

SECONDARY OUTCOMES:
Rater coding of enjoyment | One 5 minute segment per session for five months
  Trained coders rated the number of times the child expressed enjoyment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Llambias C, Magill-Evans J, Smith V, Warren S. Equine-Assisted Occupational Therapy: Increasing Engagement for Children With Autism Spectrum Disorder. Am J Occup Ther. 2016 Nov/Dec;70(6):7006220040p1-7006220040p9. doi: 10.5014/ajot.2016.020701. PMID 27767943